CLINICAL TRIAL: NCT00641563
Title: The Effects of Dexmedetomidine/Remifentanil and Midazolam/Remifentanil on Auditory-evoked Potentials and Electroencephalogram at Light-to-moderate Sedation Levels in Healthy Subjects
Brief Title: Effects of Two Different Sedation Regimes on Auditory Evoked Potentials and Electroencephalogram (EEG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Matthias Haenggi, Department of Intensive Care Medicine, university Hospital Bern - Inselspital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KIM-NMP3
Record Dates: First submitted 2008-02-25; First posted 2008-03-24 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-10

CONDITIONS: Conscious Sedation; Deep Sedation; Critical Care
Keywords: dexmedetomidine; midazolam; remifentanil; Electroencephalography; Event related potentials; BIS; Bispectral Index; Response Entropy; State Entropy
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dex/Remi followed by Mida/Remi (Active Comparator): Sedation with dexmedetomidine and remifentanil followed by sedation with midazolam and remifentanil separated by one week
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Remifentanil
- Mida/Remi followed by Dexa/Remi (Active Comparator): Sedation with midazolam and remifentanil followed by sedation with dexmedetomidine and remifentanil separated by one week
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Infusion of dexmedetomidine
Drug: Midazolam — Midazolam infusion
Drug: Remifentanil — Infusion of remifentanil

SUMMARY:
Sedation may be necessary in intensive care to facilitate diverse therapeutic interventions, but the use of sedative drugs may increase the risk of delirium and long-term cognitive impairment. Thus the implementation and monitoring of sedation remains difficult despite the use of sedation protocols and clinical sedation scores. Attempts to improve sedation monitoring through the use of the electroencephalogram(EEG) have been disappointing. Derived variables based on the unstimulated EEG fail to predict the response to external stimuli at the clinically most relevant light-to-moderate sedation levels, and the overlap between moderate and deep sedation levels is wide. We have demonstrated that long-latency auditory evoked potentials (ERPs)can be used to avoid deep levels of sedation in healthy volunteers during propofol sedation, independent of the concomitant administration of remifentanil. This approach has a potential clinical application for improved monitoring of sedation. Since the effects of different sedative drugs on the EEG may vary widely, the use of ERPs to monitor sedation needs to be evaluated with different sedative drugs. Therefore we will administer two widely used drug combinations (dexmedetomidine/remifentanil and midazolam/remifentanil) in healthy volunteers and record ERPS and processed EEG during clinical relevant sedation levels

DETAILED DESCRIPTION:
Sedation may be necessary in intensive care to facilitate diverse therapeutic interventions, but the use of sedative drugs may increase the risk of delirium and long-term cognitive impairment. Thus the implementation and monitoring of sedation remains difficult despite the use of sedation protocols and clinical sedation scores. Attempts to improve sedation monitoring through the use of the electroencephalogram (EEG) have been disappointing. Derived variables based on the unstimulated EEG fail to predict the response to external stimuli at the clinically most relevant light-to-moderate sedation levels, and the overlap between moderate and deep sedation levels is wide. We have demonstrated that long-latency auditory evoked potentials (ERPs)can be used to avoid deep levels of sedation in healthy volunteers during propofol sedation, independent of the concomitant administration of remifentanil. This approach has a potential clinical application for improved monitoring of sedation. Since the effects of different sedative drugs on the EEG may vary widely, the use of ERPs to monitor sedation needs to be evaluated with different sedative drugs. The alpha-2 agonist dexmedetomidine (dex) has been approved for short-term sedation in surgical intensive care unit (ICU) patients. Preliminary data suggest that the risk of delirium may be substantially reduced when dexmedetomidine is used to produce sedation. Since dexmedetomidine acts via different receptors and brain areas than do benzodiazepines and propofol, its impact on the brain electrophysiology may also be different. The assessment of dexmedetomidine's effects on the EEG and ERPs at various sedation levels has been limited in humans. We hypothesized that the combinations DEXMEDETOMIDINE/REMIFANTANIL (dex/remi) and MIDAZOLAM/REMIFENTANIL (mida/remi) would induce the same changes in EEG and long-latency ERPs during light-to-moderate levels of sedation in healthy subjects, despite the different quality of sedation that they provide. The opioid remifentanil was added because virtually all patients in the ICU have some level of pain and receive an opioid analgesic in combination with a sedative. 10 healthy subjects were assessed with both drug combinations (dex/remi and mida/remi), at least 7 days apart. The sequence of the drug combinations were randomized.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* healthy

Exclusion Criteria:

* History of problems during anesthesia
* Impairment of the auditory system

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2004-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Haenggi, MD, Principal Investigator — University of Bern
Locations (1):
- Departement of Intensive Care Medicine - University Hospital Bern - Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Haenggi M, Ypparila H, Takala J, Korhonen I, Luginbuhl M, Petersen-Felix S, Jakob SM. Measuring depth of sedation with auditory evoked potentials during controlled infusion of propofol and remifentanil in healthy volunteers. Anesth Analg. 2004 Dec;99(6):1728-1736. doi: 10.1213/01.ANE.0000135634.46493.0A. PMID 15562062
- [Result] Haenggi M, Ypparila H, Hauser K, Caviezel C, Korhonen I, Takala J, Jakob SM. The effects of dexmedetomidine/remifentanil and midazolam/remifentanil on auditory-evoked potentials and electroencephalogram at light-to-moderate sedation levels in healthy subjects. Anesth Analg. 2006 Nov;103(5):1163-9. doi: 10.1213/01.ane.0000237394.21087.85. PMID 17056949
- [Result] Haenggi M, Ypparila-Wolters H, Hauser K, Caviezel C, Takala J, Korhonen I, Jakob SM. Intra- and inter-individual variation of BIS-index and Entropy during controlled sedation with midazolam/remifentanil and dexmedetomidine/remifentanil in healthy volunteers: an interventional study. Crit Care. 2009;13(1):R20. doi: 10.1186/cc7723. Epub 2009 Feb 19. PMID 19228415

RESULTS

PARTICIPANT FLOW:
Groups:
- Mida/Remi Followed by Dex/Remi: Sedation with midazolam and remifentanil followed by sedation with dexmedetomidine and remifentanil separated by one week
Period: Infusion 1
Arm/Group | Dex/Remi Followed by Mida/Remi | Mida/Remi Followed by Dex/Remi
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Infusion 2
Arm/Group | Dex/Remi Followed by Mida/Remi | Mida/Remi Followed by Dex/Remi
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Both arms combined
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  Switzerland | 10

OUTCOME MEASURES:

1. Primary Outcome: Amplitudes (in Micro Volts) of Acoustic Event Related Potentials (Time-locked Amplitudes in the Electroencephalogram 100 Milliseconds After the Acoustic Stimulus, Averaged Over 40 Stimuli)Awake and at 3 Different Drug-induced Sedation Levels
Description: Event Related Potentials (time-locked amplitudes in the electroencephalogram 100 milliseconds after the acoustic stimulus, averaged over 40 stimuli) Sedation levels were graded with the Ramsay scale (RS), where the responses of patients to standardized increasing stimuli (voice, then prodding, the pain stimulus) are graded. The higher the number, the deeper is the sedation. RS 6 means no response at all (= anesthesia)
Time Frame: awake + 3 sedation levels (RS2/3/4) (20 minutes each)
Measure: Mean (Standard Deviation); unit: micro Volt
Groups:
- Dex/Remi: Sedation with dexmedetomidine and remifentanil
- Mida/Remi: Sedation with midazolam and remifentanil
Arm/Group | Dex/Remi | Mida/Remi
Number analyzed (Participants) | 10 | 10
micro Volt
  awake | -5.9 (1.3) | -5.3 (1.3)
  RS 2 | -6.4 (1.1) | -4.8 (2)
  RS 3 | -4.7 (2.4) | -2.4 (2)
  RS 4 | -3.5 (2.7) | -0.4 (1.1)

2. Secondary Outcome: BIS-Index Awake and 3 Sedation Levels (RS 2/3/4)
Description: BIS-Index is a dimensionless value ranging from 0-100, indicating fully awake at 100 and a flat-line electroencephalogram at 0. Standard anesthesia creates a BIS-Index range 40-60. The scale is ordinal, not interval. BIS Index is calculated from the EEG by a proprietary algorithm (Aspect Medical Inc.)
Time Frame: awake and 3 sedation levels (RS 2/3/4) 20 min each
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dex/Remi | Mida/Remi
Number analyzed (Participants) | 10 | 10
Units on a scale
  awake | 92.5 (4.64) | 93.7 (3.51)
  sedation level RS 2 | 84.5 (5.82) | 84.7 (5.13)
  sedation level RS 3 | 69.5 (8.05) | 73.2 (6.66)
  sedation level RS 4 | 51.4 (7.16) | 68.9 (5.70)

ADVERSE EVENTS:
Arm/Group | Dex/Remi | Mida/Remi Followed by Dex/Remi
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No